CLINICAL TRIAL: NCT01010698
Title: Evaluation of Biopharmaceutics Classification System Class 3 Drugs for Possible Biowaivers
Brief Title: Class 3 Biowaivers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, James E Polli, Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: HP-00044278; HSF223200810041C (Other Grant/Funding Number: Food and Drug Administration)
Record Dates: First submitted 2009-11-09; First posted 2009-11-10 (Estimated); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Healthy
Keywords: cimetidine; acyclovir; pharmacokinetics; excipient; formulation
MeSH Terms: interventions — Cimetidine; Acyclovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- cimetidine (or acyclovir) capsule 1 (Experimental): formulation 1
  Interventions: Drug: cimetidine (or acyclovir)
- cimetidine (or acyclovir) capsule 2 (Experimental): formulation 2
  Interventions: Drug: cimetidine (or acyclovir)
- cimetidine (or acyclovir) capsule 3 (Experimental): formulation 3
  Interventions: Drug: cimetidine (or acyclovir)
- cimetidine (or acyclovir) reference (Active Comparator): reference product
  Interventions: Drug: cimetidine (or acyclovir)

INTERVENTIONS:
Drug: cimetidine (or acyclovir) — cimetidine (or acyclovir) 200mg (single dose)

SUMMARY:
The Biopharmaceutics Classification System (BCS) is employed by the US FDA to categorize drug substances into 4 classes and to characterize drugs in terms of aqueous solubility and intestinal permeability. The four BCS categories for a drug substance are Class 1, Class 2, Class 3, and Class 4. Biopharmaceutical properties of aqueous solubility and intestinal permeability with drug product dissolution determine the rate and extent of drug absorption from immediate-release (IR) and solid oral dosages forms (e.g. tablets,capsules). Each class exhibits information regarding biopharmaceutic properties and bioequivalence. For example, Class 1 drugs have the most favorable oral biopharmaceutic properties (high solubility and high permeability). With these biopharmaceutic properties for class 1 drugs, results in vivo bioequivalence (BE) studies for rapidly dissolving IR solid oral dosage forms the FDA provided waivers. This approach alone has resulted in new and generic drugs approved based on vitro data alone (i.e. biowaived), with great savings in resources and reduction in unnecessary human testing.

Objectives: 1) The primary objective of this study is to assess whether common excipients cause bioinequivalence of Class 3 drugs. 2) The secondary objective is the results of the study will contribute towards providing scientific evidence to the FDA for consideration of Class 3 drugs for BCS-based biowaivers.

Hypotheses: The investigators anticipate that common excipients do not cause bioinequivalence. 1) Hence, the hypothesize of this study is commonly used excipients in oral medications (tablets, capsules) modulate the rate or extent of Class 3 drug absorption and result in bioinequivalence. 2) Alternative hypothesis is that commonly used excipients in oral medications (tablets, capsules) do not modulate the rate or extent of Class 3 drug absorption and do not result in bioinequivalence.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* Age 18-55
* Healthy volunteers: Subjects in good health, as determined by screening evaluation that is not greater than 30 days before the first drug study visit
* Willing to avoid caffeine containing products 24 hours prior to and day of study visits
* Willing to stop all OTC medications for 24 hours prior to and during study visits
* Able to provide informed consent

Exclusion Criteria:

* Presence of significant medical disease (including cardiovascular, pulmonary, hematologic, endocrine, immunologic, neurologic, gastrointestinal or psychiatric)
* Presence of hepatic, renal disease
* Pregnant women, breast feeding or trying to become pregnant
* Excessive alcohol use (i.e. current physical, behavioral, or personal manifestations related to the abuse or dependency on alcohol)
* Routine use (i.e. daily or weekly) prescription medication except birth control pills
* Routine use (i.e. daily or weekly) use of acid blockers, antacids, anti-diarrhea, stimulants, appetite suppressants, or anti nausea medication or other drugs that modulate GI function
* Currently taking cimetidine (or acyclovir) or medication known to interact with cimetidine (or acyclovir)
* Allergic to cimetidine (or acyclovir)
* Undergoing therapy for solid tumor or blood malignancy
* Any condition in which in the opinion of the PI or medical physician would increase risk to the subject or interfere with the integrity of the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2009-06; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Change in the amount of drug in blood during the study | 10 hours
  Plasma samples will be collected to measure level of drug

CONTACTS AND LOCATIONS:
Overall Officials: James Polli, Principal Investigator — University of Maryland, College Park
Locations (1):
- University of Maryland, Baltimore, Maryland, United States